CLINICAL TRIAL: NCT04995744
Title: Pectoralis Major Pedicle Bone Graft For 4-Part Proximal Humerus Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Bulent KARSLIOGLU, Orthopedics and Traumatology specialist, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pectoralis Major Pedicle Graft
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Patients With Closed Neer Type 4 Proximal Humerus Fractures
Keywords: proximal humerus; closed; fracture; bone pedicled graft
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with closed Neer type 4 proximal humerus fractures (Other): patients aged 50-75 years with closed Neer type 4 proximal humerus fractures
  Interventions: Procedure: Pectoralis Major Pedicle Bone Graft

INTERVENTIONS:
Procedure: Pectoralis Major Pedicle Bone Graft — It is aimed to restore the integrity of the medial cortex with the bone pedicle from the insertion region of the pectoralis major muscle in middle-aged patients with Neer type 4 proximal humerus fractures. Researchers aim to reduce the risk of avascular necrosis with a vascular living bone tissue, as well as providing mechanical support with this method. The investigators aim to reduce the risk of avascular necrosis with a vascular living bone tissue, as well as providing mechanical support with this method.

SUMMARY:
The investigators tried to evaluate the results of our patients who underwent plate osteosynthesis with vascularized pectoralis major graft for the treatment of 4-part proximal humerus fractures.

DETAILED DESCRIPTION:
The risk of avascular necrosis, nonunion, or malunion is high in 4-part fractures which is the most serious form of proximal humerus fracture.Bone impaction grafts are an important treatment option when osteosynthesis with LCP plate is desired especially for osteoporotic patients. Fibular strut grafts (FSGs) and autologous iliac bone impaction grafts (AIBIGs), which are frequently used to provide mechanical support, may have the risk of nonunion in osteoporotic bone whose vascular support is weakened due to fracture. Bone pedicled pectoralis major grafts may prevent varus collapse, nonunion and avascular necrosis.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 50-75 years with closed Neer type 4 proximal humerus fractures

Exclusion Criteria:

* Patients under 50 and over 75 years of age,
* Patients with pathological fractures,
* Patients with neurological deficits such as brachial plexus injury
* Patients with previous shoulder surgery

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Patients were evaluated in terms of functional shoulder results and radiographic union | 2 years
  Constant and American shoulder and elbow surgeons scores were used for functional assesment

CONTACTS AND LOCATIONS:
Locations (1):
- SBU Prof. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fialka C, Stampfl P, Arbes S, Reuter P, Oberleitner G, Vecsei V. Primary hemiarthroplasty in four-part fractures of the proximal humerus: randomized trial of two different implant systems. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):210-5. doi: 10.1016/j.jse.2007.07.002. Epub 2007 Oct 10. PMID 17931895
- [Result] Kim SH, Lee YH, Chung SW, Shin SH, Jang WY, Gong HS, Baek GH. Outcomes for four-part proximal humerus fractures treated with a locking compression plate and an autologous iliac bone impaction graft. Injury. 2012 Oct;43(10):1724-31. doi: 10.1016/j.injury.2012.06.029. Epub 2012 Jul 20. PMID 22819250
- [Result] Palvanen M, Kannus P, Niemi S, Parkkari J. Update in the epidemiology of proximal humeral fractures. Clin Orthop Relat Res. 2006 Jan;442:87-92. doi: 10.1097/01.blo.0000194672.79634.78. PMID 16394745
- [Result] Konrad G, Bayer J, Hepp P, Voigt C, Oestern H, Kaab M, Luo C, Plecko M, Wendt K, Kostler W, Sudkamp N. Open reduction and internal fixation of proximal humeral fractures with use of the locking proximal humerus plate. Surgical technique. J Bone Joint Surg Am. 2010 Mar;92 Suppl 1 Pt 1:85-95. doi: 10.2106/JBJS.I.01462. PMID 20194347
- [Result] Clavert P, Adam P, Bevort A, Bonnomet F, Kempf JF. Pitfalls and complications with locking plate for proximal humerus fracture. J Shoulder Elbow Surg. 2010 Jun;19(4):489-94. doi: 10.1016/j.jse.2009.09.005. Epub 2009 Dec 7. PMID 19995683
- [Result] Neer CS 2nd. Displaced proximal humeral fractures. I. Classification and evaluation. J Bone Joint Surg Am. 1970 Sep;52(6):1077-89. No abstract available. PMID 5455339
- [Result] Gallo RA, Sciulli R, Daffner RH, Altman DT, Altman GT. Defining the relationship between rotator cuff injury and proximal humerus fractures. Clin Orthop Relat Res. 2007 May;458:70-7. doi: 10.1097/BLO.0b013e31803bb400. PMID 17308477
- [Result] Choo A, Sobol G, Maltenfort M, Getz C, Abboud J. Prevalence of rotator cuff tears in operative proximal humerus fractures. Orthopedics. 2014 Nov;37(11):e968-74. doi: 10.3928/01477447-20141023-52. PMID 25361372
- [Result] Kim SH, Szabo RM, Marder RA. Epidemiology of humerus fractures in the United States: nationwide emergency department sample, 2008. Arthritis Care Res (Hoboken). 2012 Mar;64(3):407-14. doi: 10.1002/acr.21563. PMID 22162357
- [Result] Adeyemo A, Bertha N, Perry KJ, Updegrove G. Implant Selection for Proximal Humerus Fractures. Orthop Clin North Am. 2021 Apr;52(2):167-175. doi: 10.1016/j.ocl.2020.12.008. Epub 2021 Feb 10. PMID 33752838
- [Result] Hardeman F, Bollars P, Donnelly M, Bellemans J, Nijs S. Predictive factors for functional outcome and failure in angular stable osteosynthesis of the proximal humerus. Injury. 2012 Feb;43(2):153-8. doi: 10.1016/j.injury.2011.04.003. Epub 2011 May 12. PMID 21570073
- [Result] Laflamme GY, Moisan P, Chapleau J, Goulet J, Leduc S, Benoit B, Rouleau DM. Novel Technical Factors Affecting Proximal Humerus Fixation Stability. J Orthop Trauma. 2021 May 1;35(5):259-264. doi: 10.1097/BOT.0000000000001984. PMID 33165208
- [Result] Voigt C, Kreienborg S, Megatli O, Schulz AP, Lill H, Hurschler C. How does a varus deformity of the humeral head affect elevation forces and shoulder function? A biomechanical study with human shoulder specimens. J Orthop Trauma. 2011 Jul;25(7):399-405. doi: 10.1097/BOT.0b013e31820beb80. PMID 21637119
- [Result] Krappinger D, Bizzotto N, Riedmann S, Kammerlander C, Hengg C, Kralinger FS. Predicting failure after surgical fixation of proximal humerus fractures. Injury. 2011 Nov;42(11):1283-8. doi: 10.1016/j.injury.2011.01.017. Epub 2011 Feb 9. PMID 21310406
- [Result] Katthagen JC, Schwarze M, Meyer-Kobbe J, Voigt C, Hurschler C, Lill H. Biomechanical effects of calcar screws and bone block augmentation on medial support in locked plating of proximal humeral fractures. Clin Biomech (Bristol). 2014 Aug;29(7):735-41. doi: 10.1016/j.clinbiomech.2014.06.008. Epub 2014 Jun 19. PMID 24997810
- [Result] Kim YK, Kang SW, Jung KH, Oh YK. The potential of locking plate with intramedullary fibular allograft to manage proximal humeral fracture with an unstable medial column. Arch Orthop Trauma Surg. 2022 Jan;142(1):91-97. doi: 10.1007/s00402-020-03604-2. Epub 2020 Sep 18. PMID 32948917
- [Result] Gardner MJ, Weil Y, Barker JU, Kelly BT, Helfet DL, Lorich DG. The importance of medial support in locked plating of proximal humerus fractures. J Orthop Trauma. 2007 Mar;21(3):185-91. doi: 10.1097/BOT.0b013e3180333094. PMID 17473755
- [Result] McMillan TE, Johnstone AJ. Primary screw perforation or subsequent screw cut-out following proximal humerus fracture fixation using locking plates: a review of causative factors and proposed solutions. Int Orthop. 2018 Aug;42(8):1935-1942. doi: 10.1007/s00264-017-3652-6. Epub 2017 Oct 7. PMID 28988333
- [Result] Schnetzke M, Bockmeyer J, Loew M, Studier-Fischer S, Grutzner PA, Guehring T. Rate of avascular necrosis after fracture dislocations of the proximal humerus: Timing of surgery. Obere Extrem. 2018;13(4):273-278. doi: 10.1007/s11678-018-0452-6. Epub 2018 Mar 7. PMID 30546492
- [Result] Neviaser AS, Hettrich CM, Dines JS, Lorich DG. Rate of avascular necrosis following proximal humerus fractures treated with a lateral locking plate and endosteal implant. Arch Orthop Trauma Surg. 2011 Dec;131(12):1617-22. doi: 10.1007/s00402-011-1366-6. Epub 2011 Aug 4. PMID 21814772
- [Result] Peng C-H, Wu W-T, Yu T-C, Chen L-C, Hsu S-H, Kwong S-T, et al. Surgical treatment for proximal humeral fracture in elderly patients with emphasis on the use of intramedullary strut allografts. Tzu Chi Medical Journal 2012;24:131-5.
- [Result] Chen H, Ji X, Zhang Q, Liang X, Tang P. Clinical outcomes of allograft with locking compression plates for elderly four-part proximal humerus fractures. J Orthop Surg Res. 2015 Jul 22;10:114. doi: 10.1186/s13018-015-0258-9. PMID 26195025
- [Result] Reilly P, Macleod I, Macfarlane R, Windley J, Emery RJ. Dead men and radiologists don't lie: a review of cadaveric and radiological studies of rotator cuff tear prevalence. Ann R Coll Surg Engl. 2006 Mar;88(2):116-21. doi: 10.1308/003588406X94968. PMID 16551396
- [Result] Fung L, Wong B, Ravichandiran K, Agur A, Rindlisbacher T, Elmaraghy A. Three-dimensional study of pectoralis major muscle and tendon architecture. Clin Anat. 2009 May;22(4):500-8. doi: 10.1002/ca.20784. PMID 19291757
- [Result] Bois AJ, Lo IKY. Surgical anatomy of the pectoralis major tendon insertion revisited: relationship to nearby structures and the pectoral eminence for defining the anatomic footprint. JSES Int. 2020 May 7;4(2):324-332. doi: 10.1016/j.jseint.2020.02.010. eCollection 2020 Jun. PMID 32490421
- [Result] Meier JK, Spoerl S, Spanier G, Wunschel M, Gottsauner MJ, Schuderer J, Reichert TE, Ettl T. Alternatives to free flap surgery for maxillofacial reconstruction: focus on the submental island flap and the pectoralis major myocutaneous flap. BMC Oral Health. 2021 Apr 19;21(1):198. doi: 10.1186/s12903-021-01563-7. PMID 33874923
- [Result] Wyckman A, Abdelrahman I, Steinvall I, Zdolsek J, Granfeldt H, Sjoberg F, Nettelblad H, Elmasry M. Reconstruction of sternal defects after sternotomy with postoperative osteomyelitis, using a unilateral pectoralis major advancement muscle flap. Sci Rep. 2020 May 20;10(1):8380. doi: 10.1038/s41598-020-65398-y. PMID 32433505
- [Result] Aydin N, Tutuncu MN, Sekizkardes M. Pectoralis major tendon transfer for subscapularis deficiency following multiple failed instability surgeries: A case report. Acta Orthop Traumatol Turc. 2020 Nov;54(6):651-654. doi: 10.5152/j.aott.2020.19174. PMID 33424001
- [Result] Resch H, Povacz P, Maurer H, Koller H, Tauber M. Pectoralis major inverse plasty for functional reconstruction in patients with anterolateral deltoid deficiency. J Bone Joint Surg Br. 2008 Jun;90(6):757-63. doi: 10.1302/0301-620X.90B6.19804. PMID 18539669
- [Result] Freeman JL, Walker EP, Wilson JS, Shaw HJ. The vascular anatomy of the pectoralis major myocutaneous flap. Br J Plast Surg. 1981 Jan;34(1):3-10. doi: 10.1016/0007-1226(81)90086-2. PMID 7459521